CLINICAL TRIAL: NCT02075450
Title: Assessing and Improving the Quality of Cardiopulmonary Resuscitation (CPR) Delivered During Simulated Pediatric Cardiac Arrest Using a Novel Pediatric CPR Feedback Device
Brief Title: Improving the Quality of Cardiopulmonary Resuscitation (CPR) During Pediatric Cardiac Arrest
Acronym: QCPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KidSIM Simulation Program (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: E-23697
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Cardiac Arrest
Keywords: Cardiac; Arrest; Simulation; Feedback
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (No Intervention): Practice CPRcard lights not visible, Practice Just in Time Video - not provided to study participants, CPRcard lights not visible during study scenario
- Arm 2 (Experimental): Practice CPRcard light- not visible, Practice CPR Just in Time Video- not provided, CPRcard light visible during study scenario.
  Interventions: Device: CPRcard
- Arm 3 (Experimental): Practice CPRcard light- visible, Practice Just in Time Video- watched by study participant, CPRcard light- not visible during study scenario.
  Interventions: Other: Just in Time Video
- Arm # 4 (Experimental): Practice CPRcard visible and the study participants watch the Just in Time Video,CPRcard light visible during study scenario
  Interventions: Device: CPRcard; Other: Just in Time Video

INTERVENTIONS:
Device: CPRcard — CPR Card in place during chest compressions to provide immediate visual feedback.
  Other Names: CPRcard = CPR feedback device
  Arms: Arm # 4; Arm 2
Other: Just in Time Video — CPR Just in Time training video administered before the simulation case
  Arms: Arm # 4; Arm 3

SUMMARY:
Our project aims to improve the delivery and assessment of cardiopulmonary resuscitation (CPR) during pediatric cardiac arrest by introducing 2 novel approaches: 1. We will evaluate the effectiveness of a novel, credit card sized, and highly affordable "nano-card" CPR visual feedback device to improve compliance with HSFC CPR guidelines when used during simulated pediatric cardiac arrest; 2. We will also develop and study a novel, "Just-in-Time" (JIT) CPR training video, integrating proven educational methods (video-based lecture, expert modeling, practice-while-watching), and use the CPR visual feedback device to provide real-time coaching.

We hypothesize that:

H1: The use of a CPR visual feedback device will improve compliance with current HSFC CPR and resuscitation guidelines during a simulated pediatric in-hospital cardiac arrest scenario compared with standard CPR with no visual feedback.

H2: A JIT CPR Training Video, viewed by healthcare providers 2-4 weeks prior to the resuscitation event, will improve compliance with current HSFC CPR and resuscitation guidelines during simulated pediatric cardiac arrest compared with those healthcare providers with no prior exposure to the JIT CPR Training Video.

H3: That there is poor correlation between providers' perception of CPR quality and actual measured CPR quality H4: That task load varies depending on provider role and type of clinical scenario

DETAILED DESCRIPTION:
Aim 1 - To evaluate the effectiveness of a CPR visual feedback device to improve compliance with current Heart and Stork Foundation of Canada (HSFC) CPR and resuscitation guidelines during simulated pediatric cardiac arrest for a team of healthcare providers.

Aim 2 - To evaluate the effectiveness of a "Just in Time" CPR Training Video to improve compliance with current HSFC CPR and resuscitation guidelines during simulated pediatric cardiac arrest for a team of healthcare providers.

Aim 3 - To determine if there is a synergistic effect when adding Just in Time CPR Training Video with the use of the CPR visual feedback device to improve compliance with current HSFC CPR and resuscitation guidelines during a simulated pediatric cardiac arrest scenario.

Aim 4 - To determine the degree to which provider's perception of CPR quality matches actual quality of CPR

Aim 5 - To describe the task load of healthcare providers in sepsis and cardiac arrest scenarios

Participants will be recruited from ten pediatric tertiary care centers in Canada, the United States, and the United Kingdom using the methodology already piloted and studied in our existing EXPRESS investigators collaborative. Participants recruited to participate in the study will be asked to perform as members of a pediatric resuscitation team. Each team of healthcare providers will be randomized into one of four study arms. In study arm 1, resuscitation teams will participate in a simulated pediatric cardiac arrest scenario, and provide standard CPR without prior JIT training and blinded to any feedback from the CPR card during the scenario. Instead, the CPR card will be placed on the chest during compressions to collect real-time data, but the feedback lights on the card will be covered by black tape and thus, not visible to the members of the resuscitation team. In study arm 2, resuscitation teams will participate in the same scenario without prior JIT training, but provide chest compressions with the CPR card placed on the chest (and providing visual feedback) during compressions. In study arm 3, participants will be given a CPR card and asked to view the JIT training video. Following practice, they will be asked to participate in the simulated cardiac arrest scenario, and provide standard CPR without feedback from the CPR card. As in study arm 1, the CPR card will still be placed on the chest, but the feedback lights will be covered and not visible to the resuscitation team members. Finally, participants in study arm 4 will received JIT training prior to the simulated scenario, and have the CPR card in place during chest compressions to provide immediate visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* Team Member: Pediatric healthcare providers, such as nurses, nurse practitioners, and residents (pediatric emergency medicine, anesthesia, family medicine)
* Team Member: No prior experience with CPR feedback devices
* Team Member: Basic Life Support, Pediatric Advanced Life Support or Advanced Cardiac Life Support certifications within the past two years
* Team Leader: Residents (Year 2,3, or 4) in pediatrics, family medicine, anesthesia, emergency medicine training programs
* Team Leader: fellows in pediatric emergency medicine, pediatric critical care or pediatric anesthesia sub specialty training programs, attending in-patient pediatricians.
* Team Leader: No prior experience with CPR feedback devices
* Team Leader: Pediatric Advanced Life Support in the past 2 years or are Pediatric Advanced Life Support instructors

Exclusion Criteria:

* Team Member and Leader: Previous experience using, teaching with, or learning with a CPR feedback device
* Team Member and Leader: No Basic Life Support, Pediatric Advance Life Support or Adult Cardiac Life Support Certification

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Chest Compression Depth | up to 6 months
  Chest compression depth is considered shallow if <40 mm and deep if >49.99 mm. The proportion of Chest Compression with depth between 40 and 49.99 mm will be reported.

SECONDARY OUTCOMES:
Chest Compression Rate | up to 6 months
  Chest compression rates will be calculated for the entire episode. The proportion of time spent doing compressions between 90-110 compressions/min will be reported.

OTHER OUTCOMES:
No Flow Fraction | up to 6 months
  No flow time (time during cardiac arrest without chest compression delivery) will be calculated as the total scenario time minus the time with no chest compression delivery. No flow fraction (no flow fraction: proportion of cardiac arrest time without chest compression delivery) will be calculated as the no flow time divided by the total arrest time. In accordance with previous pediatric and adult CPR studies, pauses in chest compression delivery are defined as period of interruptions > 1.5 seconds.
Residual Leaning Force | up to 6 months
  Residual leaning force (grams) of delivered chest compression will be captured. The proportion of chest compression with excessive residual leaning force (>2500 grams) will be reported
Frequency of Chest Compression Switches | up to 6 months
  The number of chest compression provider switches will be recorded as the number of times there is a change in chest compression provider. A provider can be counted more than once if, in the interim, another provider has preformed chest compression of more than 1 minute before the same provider resumes compressions.
Mean difference between perceived and actual quality of CPR | up to 6 months
  As calculated by perceived performance minus actual performance, for depth and rate
Accurate estimation of CPR quality | up to 6 months
  As calculated by the absolute difference of less than 10% between perceived and actual quality of CPR, for depth and rate
NASA TLX Score | up to 6 month
  NASA TLX measures the perceived task load for healthcare providers. To be filled out by participants after each scenario

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, Study Chair — Children's Hospital of Philadelphia
Locations (11):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale University Hospital, New Haven, Connecticut
  - Children's Memorial Hospital Chicago, Chicago, Illinois
  - John Hopkins Children's Hospital, Baltimore, Maryland
  - Columbia University Hospital, New York, New York
  - Hasbro Children's Hosptial, Providence, Rhode Island
  - Children's Medical Center of Dallas, Dallas, Texas
- Canada (3):
  - Alberta Children's Hosptial, Calgary, Alberta
  - Jon Duff, Edmonton, Alberta
  - Montreal Children's Hospital, Montreal, Quebec
- Bristol Royal Hospital for Children, Bristol, Bristol, United Kingdom

REFERENCES:
- [Background] Sutton RM, Maltese MR, Niles D, French B, Nishisaki A, Arbogast KB, Donoghue A, Berg RA, Helfaer MA, Nadkarni V. Quantitative analysis of chest compression interruptions during in-hospital resuscitation of older children and adolescents. Resuscitation. 2009 Nov;80(11):1259-63. doi: 10.1016/j.resuscitation.2009.08.009. Epub 2009 Sep 4. PMID 19733427
- [Derived] Cheng A, Hunt EA, Grant D, Lin Y, Grant V, Duff JP, White ML, Peterson DT, Zhong J, Gottesman R, Sudikoff S, Doan Q, Nadkarni VM, Brown L, Overly F, Bank I, Bhanji F, Kessler D, Tofil N, Davidson J, Adler M, Bragg A, Marohn K, Robertson N, Duval-Arnould J, Wong H, Donoghue A, Chatfield J, Chime N; International Network for Simulation-based Pediatric Innovation, Research, and Education CPR Investigators. Variability in quality of chest compressions provided during simulated cardiac arrest across nine pediatric institutions. Resuscitation. 2015 Dec;97:13-9. doi: 10.1016/j.resuscitation.2015.08.024. Epub 2015 Sep 28. PMID 26417701
- [Derived] Cheng A, Brown LL, Duff JP, Davidson J, Overly F, Tofil NM, Peterson DT, White ML, Bhanji F, Bank I, Gottesman R, Adler M, Zhong J, Grant V, Grant DJ, Sudikoff SN, Marohn K, Charnovich A, Hunt EA, Kessler DO, Wong H, Robertson N, Lin Y, Doan Q, Duval-Arnould JM, Nadkarni VM; International Network for Simulation-Based Pediatric Innovation, Research, & Education (INSPIRE) CPR Investigators. Improving cardiopulmonary resuscitation with a CPR feedback device and refresher simulations (CPR CARES Study): a randomized clinical trial. JAMA Pediatr. 2015 Feb;169(2):137-44. doi: 10.1001/jamapediatrics.2014.2616. PMID 25531167